CLINICAL TRIAL: NCT06398392
Title: Radiation Dosimetry of the 18 kDa Translocator Protein Ligand [18F]PBR111 in Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prof. Daniele Zullino (Other)
Responsible Party: Sponsor-Investigator, Prof. Daniele Zullino, Professor Daniele Zullino, University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2022-00542
Record Dates: First submitted 2024-04-23; First posted 2024-05-03 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Dosimetry; Healthy
MeSH Terms: interventions — 2-(6-chloro-2-(4-(3-fluoropropoxy)phenyl)imidazo(1,2-a)pyridin-3-yl)-N,N-diethylacetamide; Positron-Emission Tomography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Drug: radiation dosimetry and biodistribution (Experimental): 6 healthy adult volunteers (3 men and 3 women) will be assigned to the radiation dosimetry group. [18F]PBR111 will be administered once.
  Interventions: Drug: [18F]PBR111; Procedure: PBR111 injection; Device: PET scan; Radiation: PBR111 dosimetry

INTERVENTIONS:
Drug: [18F]PBR111 — [18F]PBR111 is a radiotracer produced at University Hospital of Geneva in a radiopharmaceutical GMP facility. The drug product is provided as sterile solution for intravenous injection in a glass vial containing 10 mL (max) of formulated product, the maximal applicable dose being 200 MBq.
  Other Names: Preparation
Procedure: PBR111 injection — [18F]PBR111 will be administered once, intravenously in the antecubital fossa at a dose of 200 MBq
Device: PET scan — Upon administration of the radiotracer, a 120-minute PET/CT scan will be initiated.
Radiation: PBR111 dosimetry — to establish the exposure of the organs/tissues to a standard radioactive dose (200 MBq) of [18F]PBR111

SUMMARY:
The 18 kDa translocator protein (TSPO) is a mitochondrial protein that becomes overexpressed during neuroinflammatory conditions, such as in Alzheimer's disease or multiple sclerosis. TSPO is of interest because it serves as a marker for microglial and astrocytic activity, measurable via in vivo positron emission tomography (PET) molecular imaging. [18F]PBR111 is a second-generation TSPO PET radioligand with high signal specificity but a sensitivity to TSPO polymorphism, in comparison with first-generation ligands. This study focused on the biodistribution and dosimetry of [18F]PBR111 in healthy humans.

DETAILED DESCRIPTION:
This study investigated the whole-body biodistribution and radiation dosimetry of the second-generation TSPO radioligand [18F]PBR111 in healthy volunteers. The translocator protein (TSPO, 18 kDa) is a mitochondrial marker overexpressed in activated microglia and astrocytes during neuroinflammatory processes such as Alzheimer's disease, multiple sclerosis, and other neurological or systemic conditions. [18F]PBR111, a fluorine-18 labeled imidazopyridine derivative, offers high affinity and specificity for TSPO but is sensitive to the rs6971 polymorphism, leading to different binding classes (high- and mixed-affinity binders). Establishing accurate human dosimetry was essential before extending its clinical use.

Six healthy volunteers (3 females, 3 males) free from chronic or acute inflammatory, infectious, or allergic conditions were recruited under local ethics approval (Geneva University Hospitals). All participants underwent genotyping for the rs6971 polymorphism to confirm the absence of low-affinity binders. Each subject received approximately 200 MBq of [18F]PBR111 intravenously, synthesized via an automated AllInOne module using [18F]fluoride produced on an IBA 18.5 MeV cyclotron. Radiochemical preparation included QMA cartridge trapping, elution with tetrabutylammonium hydroxide, azeotropic drying, nucleophilic substitution with the precursor, purification by semi-preparative HPLC, and formulation through dual C18 SepPak cartridges, ethanol/saline elution, and sterilizing filtration. The final product was obtained with high radiochemical purity and molar activity.

Dynamic whole-body PET/CT was performed on a Siemens Biograph™ Vision 600 Edge using continuous bed motion and 10 sequential passes of increasing duration over ~130 minutes. Low-dose CT provided attenuation correction. PET images were reconstructed with OP-OSEM (2 iterations, 21 subsets), incorporating TOF and resolution modeling, and expressed as SUV (body weight normalized). Organ segmentation was achieved using a deep-learning model applied to PET/CT data, covering major target organs (liver, lungs, spleen, kidneys, red bone marrow, GI tract, urinary bladder, heart wall, pancreas, adrenals, thyroid, etc.), with the remainder of the body included for dosimetric completeness.

Organ time-activity curves were derived from decay-corrected PET data, integrated, and analyzed using OLINDA/EXM v2.2 to calculate residence times and absorbed doses. Effective dose estimates followed ICRP-103 methodology. Statistical analyses included Mann-Whitney tests (sex effects) and Friedman tests with Dunn's multiple comparisons (organ contributions).

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18 (3 male and 3 female participants)
* Fluent in French and able and willing to provide written informed consent.

Exclusion Criteria:

* Homozygosity for the rs6971 polymorphism on TSPO that results in low-affinity binding. This criterion is added because this polymorphism alters significantly the ability of the radiotracer [18F]PBR111 to bind to TSPO, hence precluding quantification.
* Absence of a stable contraceptive regimen (specifically, intrauterine contraceptive device or contraceptive treatment per os). Only women with stable contraception will be added to eliminate the risk of exposure of pregnant women and their foetus to radioactivity.
* Presence of any significant history or current diagnosis of chronic disease or syndrome (including neurological, psychiatric, cardiovascular, oncological, metabolic, rheumatological conditions).
* One or more episode(s) of acute infectious or allergic reaction in the last month before inclusion and during the study period. Again, we cannot exclude that such conditions might produce immune alterations in the brain, thus confounding the results of TSPO quantification with [18F]PBR111.
* Presence of clinically relevant laboratory abnormalities in the haematological and biochemical blood tests, as defined as laboratory values that require clinical workup and/or treatment (e.g. anaemia, hyperglycaemia, electrolyte imbalances)
* A body mass index <20 or >30 (this criterion is necessary because TSPO has been shown to be variable with respect to body mass index (113-115)).
* Exposure to research related radiation in the past five years that, when combined with this study, would place subjects above the allowable limits.
* Conditions precluding entry into the scanners (e.g. claustrophobia).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2024-06-24 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
Measurement of radiation dosimetry and biodistribution of the translocator protein radiotracer [18F]PBR111 determined with PET/CT in healthy human volunteers (3 male and 3 female participants) | 6 months
  [18F]PBR111 will be manually injected as a smooth bolus followed by a 20-ml saline flush via an intravenous catheter in the antecubital fossa placed before the scan. After injecting a standard [18F]PBR111 activity of 200 MBq, PET/CT scans will be performed on a BiographTM mCT or Vision scanner (Siemens Healthcare, Erlangen, Germany). The whole duration of the scanning protocol is about 120 minutes, consisting of CT and PET dynamic acquisitions.

SECONDARY OUTCOMES:
Calculation of the total radiation exposure of a PET/CT with 200 MBq of [18F]PBR111 | 6 months
  ROIs will be delineated manually using the Osirix software on a number of internal organs directly on the PET images with the help of the CT scan for radiation dosimetry calculations. The selected ROIs will be whole brain, left and right lung and kidney, liver, heart wall, spleen, bladder, bone marrow and organs displaying an activity concentration above background. The delineated ROIs will then be copied on all dynamic PET series to extract the time activity curves (TACs) for each organ/tissue. The total number of disintegrations (formerly referred to as residence times) will be extracted and used as input to the OLINDA/EXM software to estimate the radiation dose to organs and the effective dose to the reference adult male from mimicking the adult subjects enrolled in the study protocol.

CONTACTS AND LOCATIONS:
Locations (1):
- Geneva University Hospital, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tournier BB, Mansouri Z, Salimi Y, Ceyzeriat K, Mathoux G, Richard-Lepouriel H, Zullino D, Bois F, Zaidi H, Garibotto V, Tsartsalis S, Millet P. Radiation dosimetry of the 18 kDa translocator protein ligand [18F]PBR111 in humans. Nucl Med Biol. 2025 May-Jun;144-145:109011. doi: 10.1016/j.nucmedbio.2025.109011. Epub 2025 Mar 29. PMID 40179687